CLINICAL TRIAL: NCT00380029
Title: A Phase II Study of Erlotinib (Tarceva®) in Patients With Muscle-Invasive Bladder Cancer Undergoing Radical Cystectomy
Brief Title: Erlotinib Before and After Surgery in Treating Patients With Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: OSI Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0521; P30CA016086 (NIH)
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Erlotinib Hydrochloride; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental): erlotinib given before and after transurethral resection of a bladder tumor, TURBT
  Interventions: Drug: Erlotinib; Procedure: Radical Cystectomy

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be given at a dose of 150 mg per day for 4 weeks before undergoing planned radical cystectomy. In addition, patients will continue on erlotinib daily at a dose of 150 mg per day (qd dosing) for up to 2 years after surgery (beginning within 12 weeks of surgery) or until evidence of disease recurrence or progression
  Other Names: Tarceva
Procedure: Radical Cystectomy — Will occur 4 weeks prior to dosing with erlotinib

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving erlotinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving erlotinib after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well erlotinib works when given before and after surgery in treating patients with muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of neoadjuvant erlotinib hydrochloride on histopathological, molecular, and genetic correlates in patients undergoing radical cystectomy for muscle-invasive bladder cancer.

Secondary

* Determine the pathological complete response rate in surgical specimens from patients treated with this drug.
* Determine recurrence and progression rates after cystectomy (up to 2 years after surgery) in patients treated with neoadjuvant and adjuvant erlotinib hydrochloride.
* Determine 2- and 5-year disease-free, disease-specific, and overall survival rates in patients treated with this drug.
* Determine the safety of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive oral erlotinib hydrochloride once daily for 4 weeks. Patients then undergo radical cystectomy with curative intent. Within 12 weeks after surgery, patients resume oral erlotinib hydrochloride* once daily for up to 2 years in the absence of disease progression or unacceptable toxicity.

Note: *Patients who are candidates for adjuvant chemotherapy (e.g., found to have pathologic stage T3 (pT3), Node positive (N+) disease) do not receive erlotinib hydrochloride after surgery.

Tumor tissue is obtained at baseline (at the original or confirmatory transurethral resection of the bladder tumor) and at the time of cystectomy for analysis of drug-specific and tissue-based biomarkers by western blot, immunohistochemistry, and gene array techniques. Histopathological, molecular, and genetic correlates are analyzed to better understand the potential effects of the epidermal growth factor receptor (EGFR) inhibition in transitional cell carcinoma and to determine the effect of neoadjuvant erlotinib on gene expression. Tumor tissue is also evaluated by real-time polymerase chain reaction to confirm drug effects on expected targets and on EGFR expression, activity, and affected signaling pathways in the disease state and by microarray analysis to define expression phenotypes correlating with outcome, distinguish responders from nonresponders, and determine effects of drug treatment on gene expression in disease.

Patients are followed periodically for up to 5 years after surgery.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed muscle-invasive bladder cancer, meeting the following criteria:

  * Clinical stage T2 disease
  * No locally-extensive clinical stage T3 or T4 disease
  * No metastatic disease (N+, M+) by physical exam or radiologic evaluation
* Must have undergone prior initial or confirmatory transurethral resection of the bladder tumor (TURBT)
* Candidate for and has agreed to undergo radical cystectomy with curative intent
* No non-transitional cell carcinoma histologies

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Granulocyte count > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 times upper limit of normal
* Creatinine normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindication to erlotinib hydrochloride or other tyrosine kinase inhibitors

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or systemic chemotherapy for bladder cancer

  * Prior single-dose mitomycin C allowed at the time of TURBT
* Prior 6- or 12-week course of adjuvant intravesical Bacillus Calmette-Guerin (BCG) therapy with or without recombinant interferon alfa-2a allowed
* At least 4 weeks since other prior or concurrent radiotherapy, chemotherapy, or hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-05; Primary Completion 2010-08 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj S. Pruthi, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Pruthi RS, Nielsen M, Heathcote S, Wallen EM, Rathmell WK, Godley P, Whang Y, Fielding J, Schultz H, Grigson G, Smith A, Kim W. A phase II trial of neoadjuvant erlotinib in patients with muscle-invasive bladder cancer undergoing radical cystectomy: clinical and pathological results. BJU Int. 2010 Aug;106(3):349-54. doi: 10.1111/j.1464-410X.2009.09101.x. Epub 2010 Jan 19. PMID 20089114
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 patients were screened, 23 patients were consented to the study; three of these patients were not subsequently enrolled due to ineligibility (1) and patient decision not to enroll in the trial (2).
Period: Overall Study
Arm/Group | Erlotinib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 67.1 [61 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 20
Smoking Status [Count of Participants; unit: Participants]
  Current | 7
  Former | 10
  Never | 3

OUTCOME MEASURES:

1. Primary Outcome: EGFR Activation Signal (AKT2) Expression to Predict Sensitivity to Erlotinib
Description: Determine the effect of neoadjuvant erlotinib hydrochloride on histopathological, molecular, and genetic correlates in patients undergoing radical cystectomy for muscle-invasive bladder cancer. Gene expression of pre-treatment and post-treatment tumor samples were analyzed to define molecular determinants of response or resistance to epidermal growth factor receptor (EGFR) inhibition. Both in vitro and in vivo EGFR-associated signatures were evaluated on pre-treatment bladder tumors. Candidate molecular determinants of sensitivity to EGFR inhibition were characterized and examined for their ability to predict sensitivity to EGFR inhibitors in vitro.
Time Frame: 4 weeks before treatment and 4 weeks post treatment
Population: Only patients with tumor samples with sufficient and high quality RNA were used to generate the in vivo signatures.
Measure: Mean (Full Range); unit: fold change
Groups:
- Downstaged Tumors: transurethral resection of a bladder tumor, (TURBT) tumors resected from participants treated with neo-adjuvant erlotinib which were considered to be downstaged ( pathologic tumor stage at cystectomy <pT2 and N0)
- Not-downstaged: transurethral resection of a bladder tumor, (TURBT) tumors resected from participants treated with neo-adjuvant erlotinib which were considered to be not-downstaged ( pathologic stage at cystectomy >=pT2 or node positive (N1 or N2))
Arm/Group | Downstaged Tumors | Not-downstaged
Number analyzed (Participants) | 6 | 15
fold change | -0.29 [-0.78 to 0.04] | 0.128 [-0.61 to 0.75]

2. Secondary Outcome: Pathological Complete Response Rate
Description: Determine the pathological complete response rate (P0 rate) after undergoing radical cystectomy (RC). Evaluated using Response Evaluation Criteria In Solid Tumors (RECIST). Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 20
Participants | 5

3. Secondary Outcome: Disease Recurrence and Progression Rates After Cystectomy
Description: To determine disease recurrence/progression rates after cystectomy in patients treated with erlotinib
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 20
Participants | 4

4. Secondary Outcome: Overall Survival Rate
Description: The number of patients who remained alive and with no evidence of disease at the mean (range) follow-up of 24.8 months (3.0-36.6).
Time Frame: 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 20
Participants | 10

5. Secondary Outcome: Number of Subjects Experiencing Adverse Events
Description: The incidence of all toxicities observed during neoadjuvant and adjuvant treatment phase.Toxicity will be graded per the Common Terminology Criteria for Adverse Events (CTCAE) 2.0.
Time Frame: 4 weeks - 2 years following surgery
Population: All patients enrolled received the full 4-week neoadjuvant course of erlotinib. 12 patients continued on erlotinib in the adjuvant phase for a mean (range) duration of 29 (5-84) weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Neoadjuvant Erlotinib: erlotinib given before and after transurethral resection of a bladder tumor, TURBT
  Erlotinib: Erlotinib will be given at a dose of 150 mg per day for 4 weeks before undergoing planned radical cystectomy. Radical Cystectomy: Will occur 4 weeks prior to dosing with erlotinib
- Adjuvant Erlotinib: Patients will continue on erlotinib daily at a dose of 150 mg per day (qd dosing) for up to 2 years after surgery (beginning within 12 weeks of surgery) or until evidence of disease recurrence or progression.
Arm/Group | Neoadjuvant Erlotinib | Adjuvant Erlotinib
Number analyzed (Participants) | 20 | 12
Participants
  Rash | 15 | 6
  Anorexia | 6 | 0
  Diarrea | 6 | 1
  Fatigue | 6 | 2
  Lower urinary tract symptoms | 4 | 0
  Nausea | 3 | 0
  Cough | 3 | 2
  Dry skin | 2 | 1
  Haematuria | 2 | 0
  Vagal episode | 1 | 1
  Stomatitus | 1 | 2
  Pneumonitis | 0 | 1
  Deep vein thrombosis | 0 | 1

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 11/23
Serious Adverse Events (participants affected / at risk) | 8/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=23)
Cardiac ischemia/infarction (Cardiac disorders) | 2
Cardiovascular/Arrhythmia-Other (Abnormal EKG) (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Death NOS- Unknown cause (General disorders) | 1
Gastrointestinal-Other (Mallory-Weiss tear w/nausea, vomiting) (Gastrointestinal disorders) | 1
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 2
Infection without neutropenia (Infections and infestations) | 1
Musculoskeletal- Other (Parastomal hernia) (Musculoskeletal and connective tissue disorders) | 1
Thrombosis/embolism (Injury, poisoning and procedural complications) | 2
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=23)
Abdominal pain or cramping (Gastrointestinal disorders) | 2
Alkaline phosphatase (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Amylase (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 10
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bicarbonate (Metabolism and nutrition disorders) | 4
Bladder spasms (Renal and urinary disorders) | 1
Cardiovascular/Arrhythmia-Afib/tachycardia (Vascular disorders) | 1
Coagulation-Elevated international normalized ratio (INR) (Investigations) | 1
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
CPK (creatine phosphokinase) (Investigations) | 1
Creatinine (Investigations) | 6
Dermatology/Skin-Other (Reynaud's) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin-Other (onychomycosis -on fingers -bilaterally) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin-Other (Paronychia) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin-Other (Boils on abdomen) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin-Other (Cracked Lips) (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dizziness/lightheadedness (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Fatigue (General disorders) | 8
Gastrointestinal-Other (Gastroesophageal reflux disease) (Gastrointestinal disorders) | 1
GGT (Gamma-Glutamyl transpeptidase) (Investigations) | 2
Glaucoma (Eye disorders) | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Hematuria (in the absence of vaginal cleeding) (Renal and urinary disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 13
Hemorrhage-Other (Hemorrhoid) (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Infection with unknown ANC (Infections and infestations) | 1
Infection without neutropenia (Infections and infestations) | 3
Infection/Febrile Neutropenia-Other (Urinary tract infection - intermittent) (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Lipase (Investigations) | 1
Lymphopenia (Investigations) | 4
Mood alteration - Anxiety (Psychiatric disorders) | 1
Mood alteration - Anxiety, agitation (Psychiatric disorders) | 1
Mood alteration- Depression (Psychiatric disorders) | 3
Musculoskeletal-Other (Gout flare) (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Neuropathy-sensory (Nervous system disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain-Other (Cramping - Hands/Feet) (General disorders) | 1
Pain-Other (Pain - rash induced) (General disorders) | 1
Partial thromboplastin time (PTT) (Investigations) | 1
Platelets (Investigations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 21
Renal/Genitourinary - Other (Dysuria) (Renal and urinary disorders) | 1
Renal/Genitourinary-Other (Candida urinary tract infection (UTI)) (Renal and urinary disorders) | 1
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 3
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 1
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 2
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Taste disturbance (dysgeusia) (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 12
Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ventricular tachycardia) (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes